CLINICAL TRIAL: NCT05471453
Title: To Investigate the Effectiveness of Adjuvant Supplements Prior to in Vitro Fertilization Cycles
Brief Title: Effectiveness of Adjuvant Supplements Prior to in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Attending doctor, Department of Obstetrics and Gynecology, Principal Investigator, Assistant professor, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH21-CT8-13
Record Dates: First submitted 2022-03-08; First posted 2022-07-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Dietary Supplements
Keywords: DHEA; CoQ10; Tocotrienol; poor ovarian responder; in vitro fertilization
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DHEA group (Sham Comparator): 75 mg DHEA supplementation per day for 3 months before IVF
  Interventions: Dietary Supplement: DHEA
- DHEA+CoQ10+Tocotrienol group (Experimental): 75 mg DHEA supplementation + 30 mg CoQ10 + 300 mg Tocotrienol per day for 3 months before IVF
  Interventions: Dietary Supplement: DHEA+CoQ10+Tocotrienol
- Control group (No Intervention): No supplementation before IVF

INTERVENTIONS:
Dietary Supplement: DHEA — 75 mg DHEA supplementation per day for 3 months before IVF
  Arms: DHEA group
Dietary Supplement: DHEA+CoQ10+Tocotrienol — 75 mg DHEA supplementation + 30 mg CoQ10 + 300 mg Tocotrienol per day for 3 months before IVF
  Arms: DHEA+CoQ10+Tocotrienol group

SUMMARY:
To investigate the effect of combined DHEA, CoQ10 and tocotrienol on IVF cycles in poor ovarian responders

DETAILED DESCRIPTION:
Background There is a trend for delayed marriage and childbearing worldwide. Women undergoing in vitro fertilization (IVF) cycles are getting older. Women with advanced age are more likely to be poor ovarian responders (PORs) who have poor prognosis in IVF cycles. Numerous studies have shown that DHEA supplementation may improve IVF outcomes in PORs. Additionally, due to poor prognosis of PORs, it is quite common to combine multiple therapies instead of just one treatment. Some studies showed that CoQ10 and tocotrienol are beneficial for fertility. Thus, the aim of this study is to investigate the effect of combined DHEA, CoQ10 and tocotrienol on IVF cycles in PORs.

Objective To investigate the effect of combined DHEA, CoQ10 and Tocotrienol on PORs undergoing IVF cycles

Methods The study will be conducted from March 1st, 2022 to December 31st, 2023 in our reproductive center. We plan to enroll 120 PORs undergoing IVF cycles and divided them into four groups: (1) DHEA (n=30): 75 mg DHEA supplementation per day for three months; (2) DHEA + CoQ10 + Tocotrienol (n=30): 75 mg DHEA supplementation + 30 mg CoQ10 + 300 mg Tocotrienol per day for three months; (3) Control: no supplementation. Basic characteristics, infertility history, hormone profiles and ovarian reserve will be recorded. We will recheck serum levels of DHEA-S, FSH and AMH after DHEA supplementation. Then, during the IVF cycles, cumulus cells will be collected after oocyte retrieval to analyze genes expression and mitochondrial function. We will follow reproductive outcomes after embryo transfer.

Outcome The effect of combined DHEA, CoQ10 and Tocotrienol on cumulus cells and IVF outcomes in PORs

ELIGIBILITY:
Inclusion Criteria:

* Age 35~44
* BMI18~30 kg/m2
* Diminished ovarian reserve (AFC<5, AMH<1.2 ng/ml)

Exclusion Criteria:

* Primary ovarian insufficiency
* Congenital uterine anomaly
* Severe intrauterine adhesion
* Severe male factor
* Chromosome anomaly
* Malignancy
* Donor cycle
* having supplementation within 3 months

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | through study completion, an average of 1.75 year
  continuous presence of a fetal heartbeat over 12 weeks of a pregnancy

SECONDARY OUTCOMES:
Clinical pregnancy rate | through study completion, an average of 1.75 year
  the presence of a fetal heartbeat at 6-7 weeks of a pregnancy
mitochondrial function of cumulus cells | through study completion, an average of 1.75 year
  Oxygen consumption rate of cumulus cells

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Labrie F, Martel C, Belanger A, Pelletier G. Androgens in women are essentially made from DHEA in each peripheral tissue according to intracrinology. J Steroid Biochem Mol Biol. 2017 Apr;168:9-18. doi: 10.1016/j.jsbmb.2016.12.007. Epub 2017 Jan 30. PMID 28153489
- [Background] Lin LT, Tsui KH, Wang PH. Clinical application of dehydroepiandrosterone in reproduction: A review of the evidence. J Chin Med Assoc. 2015 Aug;78(8):446-53. doi: 10.1016/j.jcma.2014.12.008. Epub 2015 Feb 20. PMID 25708822
- [Background] Nagels HE, Rishworth JR, Siristatidis CS, Kroon B. Androgens (dehydroepiandrosterone or testosterone) for women undergoing assisted reproduction. Cochrane Database Syst Rev. 2015 Nov 26;2015(11):CD009749. doi: 10.1002/14651858.CD009749.pub2. PMID 26608695
- [Background] Zhang Y, Zhang C, Shu J, Guo J, Chang HM, Leung PCK, Sheng JZ, Huang H. Adjuvant treatment strategies in ovarian stimulation for poor responders undergoing IVF: a systematic review and network meta-analysis. Hum Reprod Update. 2020 Feb 28;26(2):247-263. doi: 10.1093/humupd/dmz046. PMID 32045470
- [Background] Xu Y, Nisenblat V, Lu C, Li R, Qiao J, Zhen X, Wang S. Pretreatment with coenzyme Q10 improves ovarian response and embryo quality in low-prognosis young women with decreased ovarian reserve: a randomized controlled trial. Reprod Biol Endocrinol. 2018 Mar 27;16(1):29. doi: 10.1186/s12958-018-0343-0. PMID 29587861
- [Background] Kamsani YS, Rajikin MH, Mohamed Nor Khan NA, Abdul Satar N, Chatterjee A. Nicotine-induced cessation of embryonic development is reversed by gamma-tocotrienol in mice. Med Sci Monit Basic Res. 2013 Mar 6;19:87-92. doi: 10.12659/MSMBR.883822. PMID 23462735
- [Background] Rajikin MH, Latif ES, Mar MR, Mat Top AG, Mokhtar NM. Deleterious effects of nicotine on the ultrastructure of oocytes: role of gamma-tocotrienol. Med Sci Monit. 2009 Dec;15(12):BR378-83. PMID 19946227
- [Background] Mohd Mutalip SS, Ab-Rahim S, Rajikin MH. Vitamin E as an Antioxidant in Female Reproductive Health. Antioxidants (Basel). 2018 Jan 26;7(2):22. doi: 10.3390/antiox7020022. PMID 29373543
- [Background] Hamirah NK, Kamsani YS, Mohamed Nor Khan NA, Ab Rahim S, Rajikin MH. Effects of Nicotine and Tocotrienol-Rich Fraction Supplementation on Cytoskeletal Structures of Murine Pre-Implantation Embryos. Med Sci Monit Basic Res. 2017 Dec 8;23:373-379. doi: 10.12659/msmbr.905447. PMID 29217815
- [Background] Abd Aziz NAA, Chatterjee A, Chatterjee R, Durairajanayagam D. Tocotrienol-rich fraction supplementation prevents foetal loss in females mated with corticosterone-treated male Sprague-Dawley rats. Andrologia. 2019 Apr;51(3):e13199. doi: 10.1111/and.13199. Epub 2018 Nov 20. PMID 30461035